CLINICAL TRIAL: NCT02120586
Title: Effects and Costs of Preventive Physiotherapy Intervention in Institutionalized Elderly People With Sarcopenia: A Randomized Controlled Trial
Brief Title: Preventive Physiotherapy Intervention in Elderly People With Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Maria dels Angels Cebria i Iranzo, PT, PhD, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1382044172319; H1382044172319 (Other: University of Valencia Research Ethics Committee)
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2017-07

CONDITIONS: Sarcopenia; Syndrome; Institutionalization
Keywords: Elderly; Institutionalization; Sarcopenia; Strength training; Muscle mass; Muscle strength; Physical performance
MeSH Terms: conditions — Sarcopenia; Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Usual care
- Respiratory training group (Experimental): Participants will breathe against a load ≥ 50% of their baseline MIP, after which loads will increase according to the participant's tolerance across the remaining training period, using a Borg scale rating of 4 to 6 on perceived exertion as an indicator of adequate training intensity.
  Intervention: Inspiratory Muscle training (12-weeks)
  Interventions: Other: Inspiratory Muscle Training (IMT).
- Peripheral training group (Experimental): Participants will load ≥ 50% of their maximum muscle force (Kg), after which load will increase according to the participant's tolerance across the remaining training period, using a Borg scale rating of 4 to 6 on perceived exertion as an indicator of adequate training intensity.
  Intervention: Peripheral muscle training (12-weeks)
  Interventions: Other: Peripheral muscle training

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT). — Supervised interval-based program consisting of seven cycles of 2-minutes work and 1-minute rest. This protocol is published as a practical guide for clinicians by Hill et al (2010).
  The sessions will take place 3 times per week over a twelve-week period for a total of 36 sessions. All participants will be familiarized with the breathing exercises over a two-week familiarization period at the beginning of the protocol. The load will be adjusted at ≥ 50% of baseline MIP. Participants remain seated in groups of 8 to 10.
  Other Names: Threshold IMT (Respironics Health Inc. Cedar Grove, NJ, USA)
  Arms: Respiratory training group
Other: Peripheral muscle training — The supervised training program consists of one cycle of 10 exercises, 12 repetitions each one. The main peripheral muscles to be trained will be those recommended by Cruz-Jentoft et al (2011): brachial biceps and triceps, pectorals, deltoid, hand flexors and extensors, spine extensor muscles, psoas-iliac, quadriceps femoris and sural triceps.
  The sessions will take place 3 times per week over a twelve-week period for a total of 36 sessions. All participants were familiarized with the force exercises over a two-week familiarization period at the beginning of the protocol. The load will be adjusted at ≥ 50% of maximum muscle force. Participants remain seated in groups of 8 to 10.
  Arms: Peripheral training group

SUMMARY:
This study evaluates two strength training protocols (one in peripheral muscles and one in inspiratory muscles) in the improvement of skeletal muscle mass and function in institutionalized elderly with sarcopenia. Participants will be assigned randomly in a control or one of both experimental groups.

DETAILED DESCRIPTION:
Sarcopenia is a syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength with a risk of adverse outcomes such as physical disability, poor quality of life and death (Goodpaster et al, 2006; Delmonico et al, 2007). The contributing factors are those related to aging process, non-optimal diet, bed rest or sedentary lifestyle, chronic diseases and certain drug treatments. Most of these factors are present in the older population with comorbidity, frequently institutionalized to receive a professional long-term care.

Since the European Working Group on Sarcopenia in Older People (Cruz-Jentoft et al, 2010) recommends using the presence of both low muscle mass and low muscle function (strength and/or physical performance) for the diagnosis of sarcopenia, interventions should be focused in both criteria. The aim of this study is to prevent loss of skeletal muscle mass and strength in institutionalized elderly with sarcopenia.

To this purpose, the investigators study undertakes two physiotherapy interventions to preventing/treating Sarcopenia, namely, maintenance of muscle mass and improvement of strength in peripheral and respiratory muscles. Both interventions are common in the following features: supervision, duration, frequency and intensity of the training program.

The primary outcomes are those related to muscle mass and strength. Secondary outcomes will be related to muscle function (muscle endurance and/or physical performance), costs and health status (number of falls and fractures, exacerbations of chronic diseases, hospitalizations and deaths during the year after concluding the physiotherapy interventions).

ELIGIBILITY:
Inclusion Criteria:

* People aged > 65 years
* Sarcopenia diagnosis (Tyrovolas et al., 2015)
* Medically stable at least 2 months before the study

Exclusion Criteria:

* Cardiorespiratory, muscular, neurological, or neuromuscular disease that could interfere in the proper performance of assessment and/or training protocols.
* Endocrine and metabolic disorders that might have had an effect on muscle mass.
* Severe disorder of hydration status that could interfere in Bioelectrical Impedance Analysis (Rubbieri et al., 2014).
* A terminal disease diagnosis.
* Mini-Mental State Examination Index ≤ 20 score.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Muscle mass | The groups will be assessed at baseline (pre-intervention) and at the end of the training program (week 12, post-intervention).
  Bioimpedance analysis (BIA) estimates the volume of fat and lean body mass. The test itself is inexpensive, easy to use, readily reproducible and appropriate for both ambulatory and bedridden patients. Reference: J Aging Phys Act 2015;23(4):597-606. Korean J Intern Med 2016;31:643-650.
Change in Maximum Respiratory Pressures (MIP and MEP) | The groups will be assessed at baseline (pre-intervention) and at the end of the training program (week 12, post-intervention).
  MIP and MEP are probably the most frequently reported non-invasive estimates of respiratory muscle strength. Ever since Black and Hyatt (1969) reported this technique it has been widely used in patients, healthy control subjects across all ages, and athletes. Pressure is recorded at the mouth during a quasi-static short (few seconds) maximal breathing. Reference: Am J Respir Crit Care Med. 2002;166:531-535.
Change in Handgrip strength | The groups will be assessed at baseline (pre-intervention) and at the end of the training program (week 12, post-intervention).
  Isometric hand grip strength is strongly related with lower extremity muscle power, knee extension torque and calf cross-sectional muscle area. In practice, there is also a linear relationship between baseline handgrip strength and incident disability for activities of daily living. Reference: Age and Aging. 2010;39:412-423.
Change in peripheral muscle strength | The groups will be assessed at baseline (pre-intervention) and at the end of the training program (week 12, post-intervention).
  Maximal isometric muscle strength (Kg) was assessed for knee extension (Quadriceps femoris) and elbow flexion (Biceps brachii). Reference: J Am Geriatr Soc 2002; 50: 461-7.

SECONDARY OUTCOMES:
Change in Maximal Voluntary Ventilation (MVV) | The groups will be assessed at baseline (pre-intervention) and at the end of the training program (week 12, post-intervention).
  This ventilatory test is a non-invasive technique and is a measure of both inspiratory and expiratory muscle endurance. The MVV is the largest volume that can be breathed in and out of the lungs during a 12 -15 second interval with maximal voluntary effort. Reference: Am J Respir Crit Care Med. 2002;166:562-564.
Change in Time performed to walk 10 m distance (10mWT). | The groups will be assessed at baseline (pre-intervention) and at the end of the training program (week 12, post-intervention).
  The 10-Meter Walk Test (10mWT) is a measure of gait speed (measurement of physical performance). The walking course consist of 14 m in a hallway: a 2 m warm-up, 10 m use for the speed measurement, and 2 m for slowing down to stop. Participants can use the assistive device (eg, cane, walker) or orthotic device (eg, ankle-foot orthosis) that they use "most often" (if any) at each time point. Reference: Phys Ther. 2010;90(2):196-208.

OTHER OUTCOMES:
Falls and fractures | Intervention costs will be recorded from the time zero to 12-weeks.
  Number of falls and resulting fractures will be checked from the medical history of participants.
Intervention costs | Intervention costs will be recorded from the time zero to 12-weeks.
  Intervention costs related to staff (supervision of training programs), consumables (Threshold IMT and weights-ballasts) and capital for intervention will be calculate in 2014 €. Reference: Rev Esp Geriatr Gerontol. 2014;49:203-209.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Cebrià i Iranzo, PT, PhD, Principal Investigator — University of Valencia; María A Tortosa Chuliá, PhD, Study Chair — University of Valencia; María J Ponce Darós, PT, PhD, Study Chair — University of Valencia; Mercè Balasch i Bernat, PT, PhD, Study Chair — University of Valencia
Locations (1):
- Grupo Gero Residencias "La Saleta", Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Results are published in a J Aging Phys Act. 2018. 1;26(4):637-646.
Supporting Information: CSR
Time Frame: 2018 Oct
Access Criteria: doi: 10.1123/japa.2017-0268
URL: https://www.ncbi.nlm.nih.gov/pubmed/29431561

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Cruz-Jentoft AJ, Triana FC, Gomez-Cabrera MC, Lopez-Soto A, Masanes F, Martin PM, Rexach JA, Hidalgo DR, Salva A, Vina J, Formiga F. [The emergent role of sarcopenia: Preliminary Report of the Observatory of Sarcopenia of the Spanish Society of Geriatrics and Gerontology]. Rev Esp Geriatr Gerontol. 2011 Mar-Apr;46(2):100-10. doi: 10.1016/j.regg.2010.11.004. Epub 2011 Jan 8. Spanish. PMID 21216498
- [Background] Doherty TJ. Invited review: Aging and sarcopenia. J Appl Physiol (1985). 2003 Oct;95(4):1717-27. doi: 10.1152/japplphysiol.00347.2003. PMID 12970377
- [Background] Tyrovolas S, Koyanagi A, Olaya B, Ayuso-Mateos JL, Miret M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM. The role of muscle mass and body fat on disability among older adults: A cross-national analysis. Exp Gerontol. 2015 Sep;69:27-35. doi: 10.1016/j.exger.2015.06.002. Epub 2015 Jun 3. PMID 26048566